CLINICAL TRIAL: NCT04328727
Title: A Non-randomized, Open Label, Multi-center, Phase II Study to Assess the Safety and Efficacy of Eltrombopag in Combination With Rabbit Anti-thymocyte Globulin (r-ATG) and Cyclosporine A (CsA) in East-Asian Patients With Treatment Naive Severe Aplastic Anemia (REACTS)
Brief Title: Combination of Eltrombopag With Immunosuppressive Therapy in East-Asian Patients With Severe Aplastic Anemia
Acronym: REACTS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CETB115G2201; 2024-000602-14 (Registry Identifier: EudraCT)
Record Dates: First submitted 2020-03-09; First posted 2020-03-31 (Actual); Results first posted 2025-07-17 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-12

CONDITIONS: Severe Aplastic Anemia (SAA)
Keywords: Treatment naïve severe aplastic anemia; SAA; eltrombopag; ETB115; immunosuppressive therapy; rabbit anti-thymocyte globulin; r-ATG; cyclosporine A; CsA; East-Asian patients
MeSH Terms: conditions — Anemia, Aplastic | interventions — eltrombopag; Antilymphocyte Serum; Cyclosporine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- eltrombopag (Experimental): Participants received eltrombopag in combination with r-ATG and CsA.
  * Eltrombopag was administered orally once daily with initial doses of 75mg/day for ≥ 12 years old and 37.5 mg/day for participants between ≥ 6 and < 12 years. Doses could be adjusted based on platelet count
  * r-ATG was administered intravenously at a dose of 2.5 to 3.5 mg/kg/day on Days 1-5
  * CsA was administered orally every 12 h at a starting dose of 3-6 mg/kg/day
  Interventions: Drug: eltrombopag; Drug: rabbit anti-thymocyte globulin (r-ATG); Drug: cyclosporine A (CsA)

INTERVENTIONS:
Drug: eltrombopag — Tablet 25mg and 12.5mg
  Other Names: ETB115
Drug: rabbit anti-thymocyte globulin (r-ATG) — r-ATG 25 mg sterile lyophilized powder in 10 mL vials for IV use
  Other Names: r-ATG
Drug: cyclosporine A (CsA) — CsA 25mg Capsule or CsA 5.0g/50mL solution for oral use
  Other Names: CsA

SUMMARY:
This study was designed to evaluate the efficacy and safety of eltrombopag when added to r-ATG and CsA in treatment naive East-Asian adult and pediatric patients with severe aplastic anemia (SAA).

DETAILED DESCRIPTION:
This was a non-randomized, open label, single arm, multi-center, Phase II study to evaluate the efficacy and safety of eltrombopag in combination with immunosuppressive therapy (IST) regimen of r-ATG + CsA in East-Asian patients with severe aplatsic anemia who had not received prior IST.

Eligible participants were enrolled into the study and received eltrombopag (from Day 1 to Week 26) concomitantly with r-ATG (on Days 1-5) and CsA (from Day 1 to Week 26) in the core treatment part.

Participants who were assessed as responders (meeting complete (CR) or partial (PR) response criteria) at Week 26 were eligible for the extension part of the study and continued treatment with eltrombopag and CsA after Week 26 up to Week 52. During the extension part, eltrombopag treatment was provided up to Week 52. CsA was maintained or tapered at the investigator's discretion according to local practice, with a total duration of at least 2 years (18 months after Week 26). There was a 30 days after end of treatment safety follow-up at the end of the extension part.

All participants were offered to enter the long term follow-up after the discontinuation of eltrombopag, with yearly efficacy and clonal evolution assessments up to Year 3 (Week 156).

ELIGIBILITY:
Inclusion Criteria:

* Written study informed consent and (where applicable) assent from the subject, parent, or guardian must be obtained prior to participation in the study.
* Subjects of East Asian ethnicity aged ≥ 6 years old at the time of written informed consent and assent form (if applicable).
* SAA characterized by:
* Bone marrow cellularity < 25%, or 25-50% with < 30% residual hematopoietic cells and pancytopenia, with at least two of the following parameters in peripheral blood:
* Absolute neutrophil count < 0.5×109/L
* Platelet count < 20×109/L
* Absolute reticulocyte count < 20×109/L
* HSCT not suitable or available as a treatment option (determined as per local practices or national guidelines), or has been refused by subject.

Exclusion Criteria:

* Prior IST with any ATG/ALG , alemtuzumab, high dose cyclophosphamide (≥ 45 mg/kg/day), CsA within 6 months, or prior thrombopoietin receptor agonists.
* Eastern Cooperative Oncology Group (ECOG) performance status (age ≥ 16 years) >2, or Lansky performance status (age < 16 years) <50.
* Prior and/or active medical history of:
* Known underlying congenital/inherited bone marrow failure or aplastic anemia (e.g.,such as but not limited to Fanconi anemia, congenital dyskeratosis, congenital amegakaryocytic thrombocytopenia, or Shwachman-Diamond Syndrome)
* Symptomatic paroxysmal nocturnal hemoglobinuria (PNH) and/or PNH clones >50% of polymorphonuclear neutrophil (PMN) or RBC at time of enrollment
* Myelodysplastic syndrome (MDS)
* Any cytogenetic abnormalities on karyotyping or FISH within 30 days of study enrollment (an evaluable karyotyping with at least 10 metaphases is mandatory for eligibility)
* Other known or suspected underlying primary immunodeficiency
* Any concomitant malignancies that have not fully recovered from treatment or have not been disease-free for 5 years
* Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) >3 times the upper limit of normal (ULN).
* Creatinine ≥ 2.5×local ULN
* Past medical history of thromboembolism within 6 months, and/or prior or current antiphospholipid antibody syndrome (APS).
* Presence of clinically active uncontrolled significant (of such severity that it would preclude the subject's ability to consent, be compliant with study procedures, tolerate protocol therapy) infection, including bacterial, fungal, mycobacterial, parasitic or viral infection, or any concurrent condition that, in the Investigator's opinion, would jeopardize the safety of the subject or compliance with the protocol
* Any severe and/or uncontrolled medical conditions which could cause unacceptable safety risks or compromise compliance with the protocol, such as:
* Known hepatocellular disease (e.g. active hepatitis or cirrhosis)
* Impairment of gastrointestinal (GI) function or gastrointestinal disease that may significantly alter the absorption of study treatment (e.g., ulcerative disease, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome)
* Active skin, mucosa, ocular or GI disorders of Grade > 1
* Presence of hepatitis B surface antigen (HBsAg) or positive hepatitis C antibody test result at screening. A positive serology for Hepatitis B (HB) is considered as a positive test for HBsAg. In addition, if serology is negative for HBsAg but hepatitis B core antibody (HBcAb) is positive (regardless of hepatitis B surface antibody (HBsAb) status), a hepatitis B virus (HBV) DNA test will be performed and if positive the patient will be excluded.
* Cardiac disorder (subjects with congestive heart disease of New York Heart Association (NYHA) functional classification Grade II/III/IV (for pediatric subjects, refer to the Grade II/III/IV of Modified ross heart failure classification for Children) should not be enrolled; subjects with NYHA Grade II due to cardiac disorder should not be enrolled but those with NYHA Grade II due to aplastic anemia (AA) may be enrolled.), arrhythmia with a risk of thrombosis (e.g. atrial fibrillation), pulmonary hypertension, or uncontrolled hypertension (>180/100 mmHg).

Ages: 6 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2020-11-04 (Actual); Primary Completion 2022-06-10 (Actual); Study Completion 2024-12-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (10):
- China (5):
  - Novartis Investigative Site, Guangzhou, Guangdong
  - Novartis Investigative Site, Zhengzhou, Henan
  - Novartis Investigative Site, Nanchang, Jiangxi
  - Novartis Investigative Site, Changchun, Jilin
  - Novartis Investigative Site, Tianjin
- Japan (3):
  - Novartis Investigative Site, Nagoya, Aichi-ken
  - Novartis Investigative Site, Fukuoka, Fukuoka
  - Novartis Investigative Site, Chuo Ku, Tokyo
- Novartis Investigative Site, Seoul, South Korea
- Novartis Investigative Site, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent expert panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data is currently available according to the process described on www.clinicalstudydatarequest.com.
URL: https://www.clinicalstudydatarequest.com

REFERENCES:
- See also: A Plain Language Trial Summary is available on www.novctrd.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=2649
- See also: A Pediatric Plain Language Trial Summary is available on www.novctrd.com — https://www.novctrd.com/ctrdweb/ppatientsummary/ppatientsummaries?periodicPatientSummaryId=700

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 12 sites in 4 different countries
Pre-assignment Details: there was an up to 30 days screening period (day -30 to -1) before first treatment (day 1).
Period: Overall Study
Arm/Group | Eltrombopag
Started (Started core part) | 36
Started extension part | 28
Started long term follow up | 34
Completed (Completed study) | 28
Not Completed | 8
Not completed — Guardian Decision | 1
Not completed — Participant decision | 4
Not completed — Death | 3

BASELINE CHARACTERISTICS:
Groups:
- Eltrombopag: Participants received eltrombopag in combination with r-ATG and CsA.
Arm/Group | Eltrombopag
Number analyzed (Participants) | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 8
  Between 18 and 65 years | 26
  >=65 years | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 34.7 (18.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 15
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 36
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Complete Response (CR) Rate at Week 26
Description: Complete response rate was defined as percentage of patients achieving complete response (CR).
  Complete response was defined as subjects meeting all the three criteria on two consecutive serial blood count measurements at least one week apart but not more than four weeks apart:
  * Absolute neutrophil count > 1.0 ×10^9/L
  * Platelet count > 100 ×10^9/L
  * Hemoglobin > 100 g/L
  The participants who discontinued from the trial before Week 26 and those that received blood products prior to response assessment (7 days prior for platelet transfusions, 14 days for RBC transfusion and 21 days for growth factors) were treated as non-responders.
Time Frame: Week 26 (6 months after starting study treatment)
Population: The Full Analysis Set (FAS) comprised of all participants to whom study treatment has been assigned and who received at least one dose of study treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Eltrombopag
Number analyzed (Participants) | 36
percentage of participants
  All participants | 16.7 [6.4 to 32.8]
  < 18 years: number analyzed (Participants) | 8
  < 18 years | 25 [3.2 to 65.1]
  18-64 years: number analyzed (Participants) | 26
  18-64 years | 15.4 [4.4 to 34.9]
  ≥ 65 years: number analyzed (Participants) | 2
  ≥ 65 years | 0 [0.0 to 84.2]

2. Secondary Outcome: Complete Response (CR) Rate
Description: as for outcome 1
Time Frame: Week 13 (3 months), Week 52 (12 months) and yearly after up to 3 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Eltrombopag
Number analyzed (Participants) | 36
percentage of participants
  Week 13 | 5.6 [0.7 to 18.7]
  Week 52 | 30.6 [16.3 to 48.1]
  Year 2 | 30.6 [16.3 to 48.1]
  Year 3 | 30.6 [16.3 to 48.1]

3. Secondary Outcome: Overall Response (ORR) Rate
Description: Overall response rate was defined as percentage of patients achieving complete response (CR) or partial response (PR).
  Partial response (PR) was defined as blood counts no longer meeting the standard criteria for severe pancytopenia in SAA, equivalent to at least 2 of the 3 criteria below, but not sufficient for a CR:
  * Absolute neutrophil count ≥ 0.5 × 10^9/L
  * Platelet count ≥ 20 × 10^9/L
  * Reticulocyte count ≥ 20 × 10^9/L
  Complete response (CR) was defined as subjects meeting all the three criteria on two consecutive serial blood count measurements at least one week apart but not more than four weeks apart:
  * Absolute neutrophil count > 1.0 ×10^9/L
  * Platelet count > 100 ×10^9/L
  * Hemoglobin > 100 g/L
Time Frame: Week 13 (3 months), 26 weeks (6 months), 52 weeks and yearly after up to 3 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Eltrombopag
Number analyzed (Participants) | 36
percentage of participants
  Week 13 | 66.7 [49.0 to 81.4]
  Week 26 | 77.8 [60.8 to 89.9]
  Week 52 | 66.7 [49.0 to 81.4]
  Year 2 | 50.0 [32.9 to 67.1]
  Year 3 | 41.7 [25.5 to 59.2]

4. Secondary Outcome: Duration of Complete Response
Description: Duration of response was derived as the time from first documented and confirmed complete response (CR) until the time of relapse or death, whichever occurred first. Duration of response was estimated using Kaplan-Meier method.
  Clinical relapse was considered as the occurrence of any of the following events in a participant who had achieved a hematological response (CR) but had subsequently lost response (not explained by any other independent concomitant medical conditions) in one blood count measurements:
  * Meeting again the criteria for SAA
  * Requirement for transfusion again for subjects who had been transfusion independent
  * Decrease in any of the peripheral blood counts to absolute neutrophil count < 0.5 x10^9/L or platelets < 20 x10^9/L.
Time Frame: Up to aproximately 3 years
Population: Participants in the Full Analysis Set (FAS) who achieved complete response. FAS comprised of all participants to whom study treatment has been assigned and who received at least one dose of study treatment.
Measure: Number (95% Confidence Interval); unit: months
Arm/Group | Eltrombopag
Number analyzed (Participants) | 11
months | NA [NA to NA] — NA: Not estimable due to insufficient number of participants with relapse or death (all participants with CR at Week 52 were still responding without any documented relapse at Year 3)

5. Secondary Outcome: Duration of Overall Response
Description: Duration of response was derived as the time from first documented and confirmed response (either CR or PR) until the time of relapse or death, whichever occurred first. Duration of response was estimated using Kaplan-Meier method.
  Clinical relapse was considered as the occurrence of any of the following events in a participant who had achieved a hematological response (CR or PR) but had subsequently lost response (not explained by any other independent concomitant medical conditions) in one blood count measurements:
  * Meeting again the criteria for SAA
  * Requirement for transfusion again for subjects who had been transfusion independent
  * Decrease in any of the peripheral blood counts to absolute neutrophil count < 0.5 x10^9/L or platelets < 20 x10^9/L.
Time Frame: Up to aproximately 3 years
Population: Participants in the Full Analysis Set (FAS) who achieved a response. FAS comprised of all participants to whom study treatment has been assigned and who received at least one dose of study treatment.
Measure: Number (95% Confidence Interval); unit: months
Arm/Group | Eltrombopag
Number analyzed (Participants) | 31
months | NA [3.1 to NA] — NA: Not estimable due to median duration of overall response not being achieved from the analysis due to insufficient number of participants with events

6. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from the date of the first dose of study treatment to the date of death due to any cause. If a subject was not known to have died, survival was censored at the date of last contact. The distribution function of OS was estimated using the Kaplan- Meier method.
Time Frame: Up to approximately 3 years
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Eltrombopag
Number analyzed (Participants) | 36
Months | NA [NA to NA] — NA: Not estimable due to median duration of overall survival being not evaluable from the Kaplan-Meyer analysis due to insufficient number of participants with events

7. Secondary Outcome: Overall Survival (OS) Rate
Description: OS was defined as the time from the date of the first dose of study treatment to the date of death due to any cause. The OS rate is the estimated probability that a patient will remain event-free up to the specified time point and was obtained from the Kaplan-Meier survival estimates. If a subject was not known to have died, survival was censored at the date of last contact.
Time Frame: Week 26, Week 52 and yearly after up to 3 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percent probability
Arm/Group | Eltrombopag
Number analyzed (Participants) | 36
percent probability
  Week 26 | 97.2 [81.9 to 99.6]
  Week 52 | 97.2 [81.9 to 99.6]
  Year 2 | 94.1 [78.3 to 95.5]
  Year 3 | 90.9 [74.4 to 97.0]

8. Secondary Outcome: Red Blood Cells (RBC) and Platelet Transfusion-free Interval Before Week 13 and 26
Description: Transfusion-free interval was defined as the time from most recent RBC/platelet transfusion preceding response assessment to the date of response assessment.
Time Frame: Week 13, 26
Population: The Full Analysis Set (FAS) subjects with response assessment at week 13 and 26. FAS comprised of all participants to whom study treatment has been assigned and who received at least one dose of study treatment.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Eltrombopag
Number analyzed (Participants) | 34
days
  RBC transfusion-free interval - Week 13 | 36.3 (25.62)
  RBC transfusion-free interval - Week 26: number analyzed (Participants) | 32
  RBC transfusion-free interval - Week 26 | 98.9 (57.97)
  Platelet transfusion-free interval - Week 13 | 34.0 (25.64)
  Platelet transfusion-free interval - Week 26: number analyzed (Participants) | 32
  Platelet transfusion-free interval - Week 26 | 97.3 (58.93)

9. Secondary Outcome: Percentage of Participants Who Become RBC Transfusion Independent
Description: Transfusion independent participants were defined as those participants who were transfusion dependent at baseline but became transfusion free for a period of ≥ 8 weeks post-baseline for RBCs.
Time Frame: From date of first dose to approximately 3 years
Population: Full Analysis Set (FAS) subjects who were transfusion dependent at baseline. FAS comprised of all participants to whom study treatment has been assigned and who received at least one dose of study treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Eltrombopag
Number analyzed (Participants) | 29
percentage of participants | 86.2

10. Secondary Outcome: Percentage of Participants Who Become Platelet Transfusion Independent
Description: Transfusion independent participants were defined as those participants who were transfusion dependent at baseline but became transfusion free for a period of ≥ 4 weeks post-baseline for platelets.
Time Frame: From date of first dose to approximately 3 years
Population: The Full Analysis Set (FAS) subjects who were transfusion dependent at baseline. FAS comprised of all participants to whom study treatment has been assigned and who received at least one dose of study treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Eltrombopag
Number analyzed (Participants) | 34
percentage of participants | 88.2

11. Secondary Outcome: Time From the Date of First Dose of Investigational Treatment to the Date of First Occurrence of Any Clonal Evolution Events
Description: Clonal evolution events were assessed by karyotyping (G-banding) and FISH (Fluorescence in situ hybridization) targeting abnormalities including, but not restricted to chromosome 3q del,5q del, monosomy 7, trisomy 8 and those associated with SAA (Severe aplastic anemia), MDS (Myelodysplastic syndrome), AML (Acute myeloid leukemia). Time to clonal evolution was to be estimated using the Kaplan-Meier method.
Time Frame: From date of first dose to approximately 3 years
Population: Participants who received at least one dose of study treatment and presented a clonal evolution event.
Measure: Number (95% Confidence Interval); unit: weeks
Arm/Group | Eltrombopag
Number analyzed (Participants) | 2
weeks | NA [NA to NA] — NA: Not estimable due to insufficient number of participants with events

12. Secondary Outcome: Plasma Pharmacokinetics (PK) Parameters of Eltrombopag: AUClast
Description: AUClast is the area under the curve from time zero to the last measurable concentration sampling time.
  Blood samples were collected from patients to assess the plasma concentrations of eltrombopag using a validated liquid chromatography - tandem mass spectrometry assay (LC-MS/MS) approach.
Time Frame: Pre-dose, and 2, 4, 6, 8 and 24 hours post-dose on Day 14 after initial dose
Population: Participants in the PAS with a an available value for the outcome measure. The Pharmacokinetic analysis set (PAS) includes all participants who received at least one dose of eltrombopag and provide at least one evaluable PK sample.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Eltrombopag
Number analyzed (Participants) | 14
ng*h/mL | 602000 (239000)

13. Secondary Outcome: Plasma Pharmacokinetics (PK) Parameters of Eltrombopag: AUCtau
Description: AUCtau is area under the curve calculated to the end of a dosing interval (tau) at steady-state
  Blood samples were collected from patients to assess the plasma concentrations of eltrombopag using a validated liquid chromatography - tandem mass spectrometry assay (LC-MS/MS) approach.
Time Frame: Pre-dose, and 2, 4, 6, 8 and 24 hours post-dose on Day 14 after initial dose
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Eltrombopag
Number analyzed (Participants) | 12
ng*h/mL | 585000 (231000)

14. Secondary Outcome: Plasma Pharmacokinetics (PK) Parameters of Eltrombopag: Ctrough
Description: Cthrough is the pre-dose concentration at the end of dose interval.
  Blood samples were collected to assess the plasma concentrations of eltrombopag using a validated liquid chromatography - tandem mass spectrometry assay (LC-MS/MS) approach.
  Eltrombopag was administered orally once daily with initial doses of 75mg/day for ≥ 12 years old and 37.5 mg/day for participants between ≥ 6 and < 12 years.
  Doses could be adjusted based on platelet count every 2 weeks by decreasing it by 25 mg/day (12.5 mg/day, for participants below 12 years old) if the platelet count was above 200×10^9/L. or interrupted if platelet count rose above 400×10^9/L. In partial response participants dose could be restarted or increased to that before the decrease if platelet counts < 30 x10^9/L, Hb< 90 g/L, ANC< 0.5 x 10^9/L or participant needed transfusion. In complete response participants dose could be restarted or increased to that before decrease if blood counts dropped to not meet CR criteria.
Time Frame: Pre-dose on day 15 after initation of eltrombopag and and pre-dose on the 15th day after each new dose up to week 26
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: ng/mL
Units Other Than Participants: measurements
Arm/Group | Eltrombopag
Number analyzed (Participants) | 26
Number analyzed (measurements) | 36
ng/mL | 20200 (9410)

15. Secondary Outcome: Plasma Pharmacokinetics (PK) Parameters of Eltrombopag: Cmax
Description: Cmax is the The maximum (peak) observed plasma drug concentration after dose administration.
  Blood samples were collected from patients to assess the plasma concentrations of eltrombopag using a validated liquid chromatography - tandem mass spectrometry assay (LC-MS/MS) approach.
Time Frame: Pre-dose, and 2, 4, 6, 8 and 24 hours post-dose on Day 14 after initial dose
Population: as for outcome 12
Measure: Median (Standard Deviation); unit: ng/mL
Arm/Group | Eltrombopag
Number analyzed (Participants) | 14
ng/mL | 32500 (12300)

16. Secondary Outcome: Plasma Pharmacokinetics (PK) Parameters of Eltrombopag: Tmax
Description: Tmax is the time to reach maximum (peak) plasma drug concentration after dose administration.
  Blood samples were collected from patients to assess the plasma concentrations of eltrombopag using a validated liquid chromatography - tandem mass spectrometry assay (LC-MS/MS) approach.
Time Frame: Pre-dose, and 2, 4, 6, 8 and 24 hours post-dose on Day 14 after initial dose
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Eltrombopag
Number analyzed (Participants) | 14
hours | 5.59 (5.64)

17. Secondary Outcome: Plasma Pharmacokinetics (PK) Parameters of Eltrombopag: CLss/F
Description: CLss/F is Apparent systemic (or total body) clearance at steady state from plasma.
  Blood samples were collected from patients to assess the plasma concentrations of eltrombopag using a validated liquid chromatography - tandem mass spectrometry assay (LC-MS/MS) approach.
Time Frame: Pre-dose, and 2, 4, 6, 8 and 24 hours post-dose on Day 14 after initial dose
Population: as for outcome 12
Measure: Mean (Standard Deviation); unit: Liter/hour
Arm/Group | Eltrombopag
Number analyzed (Participants) | 12
Liter/hour | 0.148 (0.0618)

ADVERSE EVENTS:
Time Frame: All-cause mortality: from first dose of study treatment up to 2 years after last dose including post-treatment long term follow up period up to 3.1 years approximately. Serious and Other Adverse Events: from first dose of study treatment until 30 days after last dose up to 1.1 years approximately.
Description: No adverse events where collected during the long term follow up
Groups:
- Eltrombopag (Post-treatment Long Term Follow-up): Deaths collected in the post- treatment long term follow-up period (starting from day 31 after last dose). No AEs were collected during this period
Arm/Group | Eltrombopag | Eltrombopag (Post-treatment Long Term Follow-up)
All-Cause Mortality (participants affected / at risk) | 1/36 | 2/34
Serious Adverse Events (participants affected / at risk) | 14/36 | 0/0
Other Adverse Events (participants affected / at risk) | 36/36 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Eltrombopag (N=36) | Eltrombopag (Post-treatment Long Term Follow-up) (N=0)
Drug-induced liver injury (Hepatobiliary disorders) | 1 | NA
Hepatic function abnormal (Hepatobiliary disorders) | 1 | NA
Herpes zoster (Infections and infestations) | 1 | NA
Sepsis (Infections and infestations) | 3 | NA
Urinary tract infection (Infections and infestations) | 1 | NA
Alanine aminotransferase increased (Investigations) | 1 | NA
Aspartate aminotransferase increased (Investigations) | 1 | NA
Blood bilirubin increased (Investigations) | 1 | NA
Gamma-glutamyltransferase increased (Investigations) | 1 | NA
Neutrophil count decreased (Investigations) | 1 | NA
Hyperuricaemia (Metabolism and nutrition disorders) | 4 | NA
Hypokalaemia (Metabolism and nutrition disorders) | 2 | NA
Hyponatraemia (Metabolism and nutrition disorders) | 1 | NA
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | NA
Hydronephrosis (Renal and urinary disorders) | 1 | NA
Breast hyperplasia (Reproductive system and breast disorders) | 1 | NA
Heavy menstrual bleeding (Reproductive system and breast disorders) | 1 | NA
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Eltrombopag (N=36) | Eltrombopag (Post-treatment Long Term Follow-up) (N=0)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 | NA
Cardiac failure (Cardiac disorders) | 2 | NA
Cataract (Eye disorders) | 3 | NA
Abdominal pain (Gastrointestinal disorders) | 2 | NA
Constipation (Gastrointestinal disorders) | 8 | NA
Diarrhoea (Gastrointestinal disorders) | 9 | NA
Dyspepsia (Gastrointestinal disorders) | 2 | NA
Gastrointestinal disorder (Gastrointestinal disorders) | 5 | NA
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 | NA
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | NA
Haemorrhoids (Gastrointestinal disorders) | 2 | NA
Mouth ulceration (Gastrointestinal disorders) | 6 | NA
Nausea (Gastrointestinal disorders) | 2 | NA
Stomatitis (Gastrointestinal disorders) | 5 | NA
Vomiting (Gastrointestinal disorders) | 5 | NA
Chest discomfort (General disorders and administration site conditions) | 4 | NA
Chest pain (General disorders and administration site conditions) | 2 | NA
Oedema peripheral (General disorders and administration site conditions) | 2 | NA
Pyrexia (General disorders and administration site conditions) | 12 | NA
Hepatic function abnormal (Hepatobiliary disorders) | 6 | NA
Hyperbilirubinaemia (Hepatobiliary disorders) | 11 | NA
Allergy to immunoglobulin therapy (Immune system disorders) | 2 | NA
Hypersensitivity (Immune system disorders) | 6 | NA
Immunodeficiency (Immune system disorders) | 2 | NA
Serum sickness (Immune system disorders) | 9 | NA
Cytomegalovirus infection reactivation (Infections and infestations) | 2 | NA
Infection (Infections and infestations) | 5 | NA
Neutropenic infection (Infections and infestations) | 3 | NA
Oral infection (Infections and infestations) | 2 | NA
Pneumonia (Infections and infestations) | 6 | NA
Upper respiratory tract infection (Infections and infestations) | 8 | NA
Urinary tract infection (Infections and infestations) | 2 | NA
Allergic transfusion reaction (Injury, poisoning and procedural complications) | 4 | NA
Alanine aminotransferase increased (Investigations) | 13 | NA
Aspartate aminotransferase increased (Investigations) | 3 | NA
Bilirubin conjugated increased (Investigations) | 2 | NA
Blood alkaline phosphatase increased (Investigations) | 3 | NA
Blood bilirubin increased (Investigations) | 7 | NA
Blood creatinine increased (Investigations) | 7 | NA
Blood glucose increased (Investigations) | 13 | NA
Blood pressure increased (Investigations) | 3 | NA
Blood urea increased (Investigations) | 4 | NA
Gamma-glutamyltransferase increased (Investigations) | 10 | NA
Decreased appetite (Metabolism and nutrition disorders) | 3 | NA
Fluid retention (Metabolism and nutrition disorders) | 9 | NA
Hypercholesterolaemia (Metabolism and nutrition disorders) | 2 | NA
Hyperglycaemia (Metabolism and nutrition disorders) | 6 | NA
Hyperlipidaemia (Metabolism and nutrition disorders) | 4 | NA
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 6 | NA
Hyperuricaemia (Metabolism and nutrition disorders) | 14 | NA
Hypoalbuminaemia (Metabolism and nutrition disorders) | 10 | NA
Hypocalcaemia (Metabolism and nutrition disorders) | 2 | NA
Hypokalaemia (Metabolism and nutrition disorders) | 18 | NA
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 | NA
Hyponatraemia (Metabolism and nutrition disorders) | 5 | NA
Hypoproteinaemia (Metabolism and nutrition disorders) | 4 | NA
Sodium retention (Metabolism and nutrition disorders) | 3 | NA
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | NA
Dizziness (Nervous system disorders) | 2 | NA
Headache (Nervous system disorders) | 4 | NA
Acute kidney injury (Renal and urinary disorders) | 3 | NA
Renal failure (Renal and urinary disorders) | 2 | NA
Renal impairment (Renal and urinary disorders) | 5 | NA
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2 | NA
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 2 | NA
Acne (Skin and subcutaneous tissue disorders) | 2 | NA
Dry skin (Skin and subcutaneous tissue disorders) | 2 | NA
Rash (Skin and subcutaneous tissue disorders) | 7 | NA
Hypertension (Vascular disorders) | 7 | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2021-12-22): https://cdn.clinicaltrials.gov/large-docs/27/NCT04328727/Prot_000.pdf
  • Statistical Analysis Plan (2024-11-11): https://cdn.clinicaltrials.gov/large-docs/27/NCT04328727/SAP_001.pdf